CLINICAL TRIAL: NCT06489171
Title: Oncological and Obstetrical Outcomes for Fertility Preservation in Early Cervical Cancer Patient With Laparoscopic-assisted Vaginal Radical Trachelectomy
Brief Title: Research on Laparoscopic Fertility-Sparing Surgery in Early-Stage Cervical Cancer
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: S-K789
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Received laparoscopic-assisted vaginal radical trachelectomy — The LAVRT procedure began with laparoscopic pelvic lymphadenectomy, and all lymph nodes were removed for frozen pathological analysis. The laparoscopic-assisted vaginal radical trachelectomy procedure was continued only if the nodes were negative. The pararectal pouch was revealed, and the uterine arteries were divided from their origin to the internal iliac artery. The ureters were freed from the posterior leaf of the broad ligament down to the level where they entered the ureteral tunnel and then displaced laterally. The uterosacral ligaments, cardinal ligaments, and parametrial portions were then divided and dissected. The section of the procedure was performed laparoscopically. The vaginal epithelium was circumferentially incised approximately 3 cm distal to the endocervix. Frozen section analysis confirmed no cancer involvement at the endocervical or vaginal margin. The vaginal mucosa was sutured to the cervical stump to form a "new cervical os".

SUMMARY:
Purpose: To evaluate the oncological and obstetrical outcomes of women with early-stage cervical cancer who underwent laparoscopic-assisted vaginal radical trachelectomy (LAVRT). All women with early-stage cervical cancer who planned to undergo fertility-preserved radical trachelectomy. The obstetric outcome evaluation was restricted to women with ≥12 months of follow-up and an active desire to conceive. The oncological outcome was evaluated in all patients.

Statistical methods: Statistical analyses were performed using IBM SPSS Statistics, version 26. The t-test is used for analyzing the continuous variables and the chi-squared test for categorical variables.

DETAILED DESCRIPTION:
This retrospective cohort study reported the reproductive intentions and outcomes of cervical cancer patients who underwent laparoscopic-assisted vaginal radical trachelectomy (LAVRT) .The LAVRT procedure began with laparoscopic pelvic lymphadenectomy, and all lymph nodes were removed for frozen pathological analysis. The laparoscopic-assisted vaginal radical trachelectomy procedure was continued only if the nodes were negative. The pararectal pouch was revealed, and the uterine arteries were divided from their origin to the internal iliac artery. The ureters were freed from the posterior leaf of the broad ligament down to the level where they entered the ureteral tunnel and then displaced laterally. The uterosacral ligaments, cardinal ligaments, and parametrial portions were then divided and dissected. The section of the procedure was performed laparoscopically. The vaginal epithelium was circumferentially incised approximately 3 cm distal to the endocervix. Frozen section analysis confirmed no cancer involvement at the endocervical or vaginal margin. The vaginal mucosa was sutured to the cervical stump to form a "new cervical os".

Postoperative adjuvant chemotherapy is indicated when women have at least one of 3 intermediate risk factors: stromal invasion of more than half of the cervix, lymphovascular space invasion (LVSI), or a tumor diameter of 4 cm or greater. Platinum-based chemotherapy (combination of paclitaxel and cisplatin or carboplatin for 3 courses) was used for these women.

Women attended follow-up visits every 3 months for the first 2 years, every 6 months for the next 3 years, and annually every year thereafter. At each follow-up visit, a physical and gynecological examination and a conventional Pap smear combined with an HPV test were performed. Abdominal (including both kidneys) and pelvic ultrasound (US) and serum tumor marker (SCC antigen or CA125 for adenocarcinoma) data were also included.

When tumor recurrence was suspected based on clinical findings or imaging studies, a positron emission tomography (PET)-CT scan was performed to investigate the extent of disease. Recurrence was confirmed by a lesion on biopsy or a positive PET-CT scan. The follow-up duration was measured from the day of the operation to the day of the last follow-up, death or loss to follow-up.

ELIGIBILITY:
Inclusion Criteria:

* (i) were younger than 45 years old; (ii) strong desired to preserve fertility; (iii) had International Federation of Gynecology and Obstetrics (FIGO) stage IA1 (with lymphovascular space invasion (LVSI) positivity) to IB2; (iv) pathologically confirmed invasive cervical cancer; (v)had histology indicative of squamous cell carcinoma, adenosquamous cancer or adenocarcinoma; (vi) lacked evidence of pelvic lymph node or distant metastasis according to pelvic MRI and serum tumor markers (SCC and CA125) levels.

Exclusion Criteria:

* (i) diagnosis of cervical gastric adenocarcinoma, cervical neuroendocrine carcinoma and other special types; (ii) invasion of cervical internal orifice; (iii) had contraindication of pregnancy; (iv) incomplete clinical data; (v) radiotherapy or hysterectomy was performed after diagnostic conization.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study will include 132 patients with early-stage cervical cancer, who undergo laparoscopic-assisted vaginal radical trachelectomy.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2003-01-01 (Actual); Primary Completion 2013-01-01 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival | 5-10 years
  the date of the treatment to the date of disease progression or death from any cause in the absence of progression
Pregnancy rate after surgery | 5 years
  Postoperative patients who have successfully conceived
Recurrence rate | 20years
  The ratio of recurrent patients to the total enrolled patients

SECONDARY OUTCOMES:
Average operation time | Intraoperative
  The length of the surgery
bleeding volume | Intraoperative
  the amount of blood loss in the patient

REFERENCES:
- [Background] Kyrgiou M, Mitra A, Paraskevaidis E. Fertility and Early Pregnancy Outcomes Following Conservative Treatment for Cervical Intraepithelial Neoplasia and Early Cervical Cancer. JAMA Oncol. 2016 Nov 1;2(11):1496-1498. doi: 10.1001/jamaoncol.2016.1839. PMID 27356074
- [Background] Martinelli F, Ditto A, Filippi F, Vinti D, Bogani G, Leone Roberti Maggiore U, Evangelista M, Signorelli M, Chiappa V, Lopez S, Somigliana E, Raspagliesi F. Conization and lymph node evaluation as a fertility-sparing treatment for early stage cervical cancer. Int J Gynecol Cancer. 2021 Mar;31(3):457-461. doi: 10.1136/ijgc-2020-001740. PMID 33649014
- [Background] Kyrgiou M, Athanasiou A, Arbyn M, Lax SF, Raspollini MR, Nieminen P, Carcopino X, Bornstein J, Gultekin M, Paraskevaidis E. Terminology for cone dimensions after local conservative treatment for cervical intraepithelial neoplasia and early invasive cervical cancer: 2022 consensus recommendations from ESGO, EFC, IFCPC, and ESP. Lancet Oncol. 2022 Aug;23(8):e385-e392. doi: 10.1016/S1470-2045(22)00191-7. PMID 35901834
- [Background] Fokom Domgue J, Schmeler KM. Conservative management of cervical cancer: Current status and obstetrical implications. Best Pract Res Clin Obstet Gynaecol. 2019 Feb;55:79-92. doi: 10.1016/j.bpobgyn.2018.06.009. Epub 2018 Jun 28. PMID 30029960
- [Result] Cao DY, Yang JX, Wu XH, Chen YL, Li L, Liu KJ, Cui MH, Xie X, Wu YM, Kong BH, Zhu GH, Xiang Y, Lang JH, Shen K; China Gynecologic Oncology Group. Comparisons of vaginal and abdominal radical trachelectomy for early-stage cervical cancer: preliminary results of a multi-center research in China. Br J Cancer. 2013 Nov 26;109(11):2778-82. doi: 10.1038/bjc.2013.656. Epub 2013 Oct 29. PMID 24169350